CLINICAL TRIAL: NCT01854671
Title: Investigating the Effect of a Prenatal Family Planning Counseling Intervention Led by Community Health Workers on Postpartum Contraceptive Use Among Women in the West Bank
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood League of Massachusetts (Other)
Collaborators: Society for Family Planning Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: SFPRF13-10
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Focus: Contraceptive Counseling; Focus: Postpartum Contraception
Keywords: postpartum contraception; contraceptive counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard care (No Intervention)
- family planning counseling led by community health worker (Experimental): The family planning counseling sessions led by community health workers will present advantages of birth spacing, available methods of postpartum contraception, contraindications (if any) for the method, when each method can be safely started postpartum, where each method can be obtained, and importance of 6 week postpartum clinic follow-up. There will also be a take-home contraceptive method brochure given at conclusion of information session -primarily pictorial and in Arabic, to facilitate discussion at home with husbands and family members.
  Interventions: Other: family planning counseling let by community health workers

INTERVENTIONS:
Other: family planning counseling let by community health workers — The family planning counseling sessions led by community health workers will present advantages of birth spacing, available methods of postpartum contraception, contraindications (if any) for the method, when each method can be safely started postpartum, where each method can be obtained, and importance of 6 week postpartum clinic follow-up. There will also be a take-home contraceptive method brochure given at conclusion of information session -primarily pictorial and in Arabic, to facilitate discussion at home with husbands and family members.
  Arms: family planning counseling led by community health worker

SUMMARY:
The purpose of this study is to measure the difference in proportion of postpartum women using contraception after a Community Health Worker (CHW) family planning educational intervention compared to women who receive standard care in the West Bank district of Ramallah and Al-Bireh.

Primary hypothesis: Postpartum contraceptive use will increase in women who receive a dedicated family planning counseling intervention delivered by CHWs during antenatal care compared to women receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* Women attending the MoH Ramallah or Al-Bireh clinic for antenatal care and 34-38 weeks pregnant at enrollment
* Planning delivery at an MoH hospital
* Able and willing to be contacted by phone or home visit

Exclusion Criteria:

* Women less than 34 weeks pregnant or non-pregnant
* Planning delivery at a private or NGO hospital
* Unwilling to be contacted for follow-up after enrollment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Self-reported contraceptive use | 6 months post-partum

SECONDARY OUTCOMES:
Intent to use contraception in the future | 6 months postpartum
Non-desire to use contraception | 6 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, MD, MPH, Principal Investigator — Planned Parenthood League of Massachusetts
Locations (1):
- Palestinian Ministry of Health Maternal Child Health Clinics (Ramallah and Al-Bireh), Ramallah and Al-Bireh, West Bank, Palestinian Territories